CLINICAL TRIAL: NCT03507075
Title: Remote Alcohol Monitoring to Facilitate Abstinence Reinforcement: Feasibility
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mikhail Koffarnus (Other)
Responsible Party: Sponsor-Investigator, Mikhail Koffarnus, Research Assistant Professor, Virginia Polytechnic Institute and State University
Organization: Virginia Polytechnic Institute and State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AA022727 (NIH)
Record Dates: First submitted 2018-04-07; First posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingent (Active Comparator): The Contingent group will receive nearly immediate monetary payments over the internet each day they remotely provide negative breathalyzer samples, but will not receive the payments if they provide positive samples or fail to provide samples in a timely manner.
  Interventions: Behavioral: Contingency management: Contingent incentives
- Noncontingent (Sham Comparator): The Noncontingent group will receive payments each day they successfully provide samples independent of the alcohol content of those samples.
  Interventions: Behavioral: Contingency management: Noncontingent incentives

INTERVENTIONS:
Behavioral: Contingency management: Contingent incentives — Monetary incentives are delivered to participants contingent upon on-time breathalyzer submissions and verified abstinence from alcohol.
  Arms: Contingent
Behavioral: Contingency management: Noncontingent incentives — Monetary incentives are delivered to participants contingent upon on-time breathalyzer submissions only with no contingency on alcohol use.
  Arms: Noncontingent

SUMMARY:
Directly reinforcing abstinence from alcohol with monetary incentives is an effective treatment for alcohol dependence, but barriers in obtaining frequent, verified biochemical measures of abstinence limit the dissemination of this treatment approach. The goal of this feasibility study is to determine if using technological advancements to remotely, accurately, and securely monitor alcohol use with a newly developed breathalyzer is an effective treatment that is acceptable to participants. If validated, this treatment approach has the potential to facilitate the dissemination of an effective, evidence-based treatment for alcohol dependence to a broader population whose treatment needs are not currently being adequately met.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Provide written informed consent
* Meet Diagnostic and Statistical Manual criteria for alcohol use disorder
* Express a desire to cut down or quit drinking

Exclusion Criteria:

* Pregnant or lactating
* Meet Diagnostic and Statistical Manual criteria for other substance use disorder (except caffeine or nicotine)
* Score 23 or greater on the Alcohol Withdrawal Symptom Checklist
* Have immediate plans to move out of the area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-11-15 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-01-05 (Actual)

PRIMARY OUTCOMES:
Percent days abstinent from alcohol during intervention | Percent days abstinent is the aggregate measure throughout the 21-day intervention period
  Three breathalyzer assessments will be collected per day during the treatment period. This outcome measure will consist of the percent days when all three breathalyzers were on time and negative for alcohol.
Treatment acceptability | Baseline, one day after treatment end, and at a one-month follow-up
  Participant ratings of treatment acceptability will be collected during assessment sessions

IPD SHARING:
Plan to Share IPD: Yes
Final research data for this project will be made as available as possible, while safeguarding the privacy of participants and protecting all confidential and proprietary data. Data will be available for use after the main findings from the final dataset have been accepted for publication. The data and associated documentation will only be made available to users under a Data Use Agreement that provides for 1) a commitment to using the data only for research purposes and not to identify any individual participant and 2) a commitment to destroying or returning the data after analyses are completed. To ensure compliance with HIPAA regulations, only a Limited Data Set will be available for use. The method of data release will be determined on a case-by-case basis depending upon the amount and type of data required.
Supporting Information: Study Protocol, SAP, ICF